CLINICAL TRIAL: NCT07312097
Title: Could Conservative Treatment Become the New Gold Standard in the Treatment of Acute Achilles Tendon Ruptures: A Prospective Randomized Controlled Trial
Brief Title: Could Conservative Treatment Become the New Gold Standard in Achilles Tendon Ruptures?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 113-2023
Record Dates: First submitted 2025-12-01; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Acute Achilles Tendon Rupture
Keywords: achilles tendon rupture; Isokinetic strength; Functional rehabilitation; conservative treatment
MeSH Terms: interventions — Conservative Treatment; Wound Healing

STUDY DESIGN:
Intervention Model Description: Participants were allocated in a 1:1 ratio to either the conservative treatment group or the surgical repair group using a parallel assignment model. Both groups received standardized early functional rehabilitation protocols specific to their treatment type, and outcomes were compared after a minimum 12-month follow-up.
Masking Description: No parties were masked in this trial. Both participants and investigators were aware of the assigned treatment group throughout the study. Outcome assessments were performed openly, without blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conservative Treatment (Active Comparator): Participants follow the GAPNOT functional rehabilitation protocol, including initial immobilization in plantar flexion, gradual partial to full weight-bearing, and supervised physiotherapy to improve plantar flexion strength and ankle range of motion.
  Interventions: Other: Conservative treatment
- Surgical Repair (Active Comparator): Open end-to-end Achilles tendon repair using the locked Krackow suture technique, followed by epitendinous augmentation and standardized early functional rehabilitation including gradual weight-bearing and physiotherapy.
  Interventions: Procedure: Surgical Repair

INTERVENTIONS:
Other: Conservative treatment — Participants follow the GAPNOT functional rehabilitation protocol. Initially immobilized in maximum plantar flexion with non-weight-bearing. At 2 weeks partial weight-bearing is allowed with an Achilles boot and heel lifts; by weeks 4-6 weight-bearing is increased and supervised physiotherapy is initiated focusing on plantar flexion strength, calf strengthening and ankle range of motion. Outcomes assessed at 12-18 months by isokinetic testing and clinical scores.
  Arms: Conservative Treatment
Procedure: Surgical Repair — Participants undergo open end-to-end Achilles tendon repair using the locked Krackow suture technique with 2-0 FiberWire and epitendinous augmentation. Postoperatively, standardized early functional rehabilitation is applied including gradual weight-bearing, ankle mobilization and physiotherapy focused on plantar flexion strength and ROM. Outcomes assessed at 12-18 months by isokinetic testing and clinical scores.
  Arms: Surgical Repair

SUMMARY:
This study aims to compare conservative and surgical treatments for acute Achilles tendon rupture. Forty-four patients were randomly assigned to either a conservative rehabilitation protocol or open surgical repair. Functional outcomes were evaluated using isokinetic muscle strength testing and clinical scoring systems such as the ATRS, AOFAS, FADI, VAS, and Leppilahti scores.

The results showed no significant difference between the two groups in terms of strength, tendon length, or clinical outcomes. Rerupture rates were similar, while wound complications occurred only in the surgical group.

The findings suggest that conservative treatment combined with early functional rehabilitation can provide outcomes comparable to surgery, with fewer complications. Conservative treatment may be a safe and effective alternative for managing acute Achilles tendon ruptures.

DETAILED DESCRIPTION:
Achilles tendon rupture is a common sports-related injury, and the optimal treatment approach remains controversial. Surgical repair has traditionally been considered the gold standard due to lower rerupture rates and better restoration of tendon continuity. However, surgery carries risks such as wound infection, nerve injury, and postoperative complications.

Recent advances in rehabilitation techniques have led to renewed interest in conservative management, which allows for early mobilization and functional recovery without surgical risks. This study was designed as a prospective, randomized clinical trial to objectively compare conservative and surgical treatments for acute Achilles tendon rupture.

Forty-four patients were randomly allocated to either a conservative treatment protocol based on the GAPNOT early functional rehabilitation model or open surgical repair using the Krackow suture technique. Functional recovery was assessed using isokinetic muscle testing for plantar flexion and dorsiflexion strength, as well as validated clinical scoring systems (ATRS, AOFAS, FADI, VAS, and Leppilahti).

The primary objective of this study is to determine whether conservative treatment can achieve comparable functional and biomechanical outcomes to surgical repair while minimizing complications. The results are expected to contribute to establishing evidence-based treatment guidelines and may support conservative management as a new gold standard in selected patient populations.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-50 years
* Acute complete Achilles tendon rupture (tendon-to-tendon)
* Injury occurred within 3 weeks prior to presentation
* Willingness and ability to comply with the functional rehabilitation program

Exclusion Criteria:

* Injury occurred more than 3 weeks prior to presentation
* Open Achilles tendon rupture
* History of preexisting foot or ankle pathology
* Musculotendinous, insertional, or calcaneal avulsion-type Achilles tendon injuries
* Presence of additional risk factors increasing Achilles tendon injury risk (e.g., diabetes mellitus, immunosuppressive therapy, fluoroquinolone use, or systemic corticosteroid use)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-08-20 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Peak Plantar Flexion Torque | 12-18 months post-injury
  Peak plantar flexion torque (Newton-meters, Nm) measured using an isokinetic dynamometer (HUMAC NORM 2015) at a standardized angular velocity.
Total Work During Plantar Flexion | 12-18 months post-injury
  Total work during plantar flexion (Joules) measured using an isokinetic dynamometer (HUMAC NORM 2015) at a standardized angular velocity.
Initial Plantar Flexion Torque | 12-18 months post-injury
  Initial plantar flexion torque (Newton-meters, Nm) measured using an isokinetic dynamometer (HUMAC NORM 2015) at a standardized angular velocity

SECONDARY OUTCOMES:
Achilles Tendon Resting Angle (ATRA) | 12-18 months post-injury
  Achilles tendon resting angle (degrees) measured using a standardized clinical goniometric method.
Pain Intensity (VAS) | 12-18 months post-injury
  Pain intensity measured using the Visual Analog Scale (VAS), reported on a 0-10 scale
Leppilahti Achilles tendon rupture score | 12-18 months post-injury
  Leppilahti Achilles tendon rupture score (points) measured using the standardized Leppilahti scoring system.
American Orthopaedic Foot and Ankle Society (AOFAS) hindfoot score | 12-18 months post-injury
  American Orthopaedic Foot and Ankle Society (AOFAS) hindfoot score (points) measured using the standardized AOFAS scoring system
Foot and Ankle Disability Index (FADI) | 12-18 months post-injury
  Foot and ankle function measured using the Foot and Ankle Disability Index (FADI), reported as a numerical score (points)
Rerupture Rate | 12-18 months post-injury
  Achilles tendon rerupture determined by clinical examination and/or imaging confirmation and recorded as the number of participants experiencing rerupture.

CONTACTS AND LOCATIONS:
Locations (1):
- Haseki Training and Research Hospital, Istanbul, Haseki Training and Research Hospital, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. The decision is based on patient confidentiality, ethical considerations, and the study's informed consent process, which did not include provisions for data sharing with external researchers

REFERENCES:
- See also: Official website of Haseki Training and Research Hospital, where the study on conservative versus operative treatment of acute Achilles tendon rupture was conducted. Provides hospital information and contact details for study-related queries. — https://hasekieah.saglik.gov.tr